CLINICAL TRIAL: NCT02368496
Title: Parenteral Nutrition and Bone Trophicity
Brief Title: APOSTrophe Study (Parenteral Nutrition and Bone Trophicity) Impact of a Long-term Parenteral Nutrition on Bone Metabolism Measured by High Resolution Peripheral Quantitative Computer Tomography (HR-pQCT) in Children and Young Adults
Acronym: APOSTROPHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013.825; 2013-A01245-40 (Other: (N°ID-RCB) France: Agence Nationale de Sécurité du Médicament et des produits de santé)
Record Dates: First submitted 2014-07-15; First posted 2015-02-23 (Estimated); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Long-term Parenteral Nutrition (2 Years) in Children and Adults
Keywords: Long-term parenteral nutrition; HR-pQCT; DXA; Bone trophicity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Children and young adults on long-term parenteral nutrition (Experimental): long-term parenteral nutrition : 2 years
  Interventions: Device: HR-pQCT

INTERVENTIONS:
Device: HR-pQCT

SUMMARY:
Recent progress in parenteral nutrition has contributed to improve vital prognosis and to reduce morbidity in patients with severe intestinal failure.

Currently, home parenteral nutrition is the only alternative to prolonged hospitalization for those patients. However, long-term parenteral nutrition can result in complications especially in bone, such as osteopenia or osteomalacia, then increasing the risk of fractures. Children are especially at risk because of bone growth and peak mineralization acquisition during puberty.

Moreover, frequency and risk factors of those complications are not well documented for children.

Dual-energy X-ray Absorptiometry (DXA) is considered as the golden standard for bone mineralization measurement. In pediatrics, this technique has some limits such as the underestimation of Bone Mineral Density (BMD) in short stature, the overestimation of the BMD in tall children, and the inability to distinguish cortical from trabecular bone or to evaluate the bone microarchitecture.

HR-pQCT, High Resolution peripheral Quantitative Computed Tomography enables noninvasive assessment of bone microarchitecture (virtual bone biopsy) using a radiation similar to DXA. However this technique has never been validated in patients with long-term parenteral nutrition.

During the usual follow-up of the patients, HR-pQCT will be the only exam which will come in addition to the routine medical tests.

ELIGIBILITY:
Inclusion Criteria:

* Patient who's receiving a long-term parenteral nutrition (over 2 years)
* Patient between 9 and 30 years of age (children big enough to stay immobile for 3 min during the measurement)
* Affiliation to the Social Security System
* Informed consent form signed by parents and assent given by the patient

Exclusion Criteria:

* Patient presenting a bone disease which is not directly related to the parenteral nutrition.
* Long-term corticotherapy ( over 6 months of therapy)
* Inability to keep the leg or the arm immobile for 3 min
* Patient not affiliated to a Social Security System
* Patient participating to another interventional study
* Pregnant patient or patient who desires pregnancy
* All situation that the physician estimated that is not compatible with the study

Ages: 9 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2014-03; Primary Completion 2015-08 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Bone mineral density (BMD) and Bone mineral contain (BMC) height z-score at baseline | J0 (baseline)
  BMD and BMC z scores (after correction for the height) will be measured by High Resolution peripheral Quantitative Computed Tomography (HR-pQCT) and compared to those measured in a control group (healthy subjects matched on age and sex). The same measurements will be also compared with those obtained by Dual-energy X Ray (DXA) but in this case each subject will be considered as his own control.

SECONDARY OUTCOMES:
Trabecular and cortical BMD z score | J0 (baseline)
  Trabecular and cortical BMD (height) z score measured by HR-pQCT for patients under parenteral nutrition at baseline will be compared to those of the control group
BMD and BMC height z score after 1 year of parenteral nutrition (PN) | 1 year
  BMD and BMC (height) z score measured by HR-pQCT and DXA after one year of PN will be compared, for each subject, to the measurements recorded at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Noel Peretti, Dr, Principal Investigator — Hospices Civils de Lyon - Hôpital Femme Mère Enfant
Locations (2):
- France (2):
  - Hospices Civils de Lyon - Hôpital Femme Mère Enfant, Bron
  - Hospices Civils de Lyon - Hôpital de la Croix-Rousse, Lyon

REFERENCES:
- [Result] Louazon T, Poinsot P, Restier L, Belmalih A, Loras-Duclaux I, Marotte S, Heissat S, Barnoud D, Chambrier C, Confavreux CB, Lachaux A, Bacchetta J, Peretti N. A prospective case-control pilot study to evaluate bone microarchitecture in children and teenagers on long-term parenteral nutrition using HR-pQCT. Sci Rep. 2021 Apr 28;11(1):9151. doi: 10.1038/s41598-021-88366-6. PMID 33911128